CLINICAL TRIAL: NCT04142762
Title: A Phase 1, Open-Label, Fixed-Sequence Study to Evaluate CYP3A4-Mediated, Oral Contraceptive, and pH Modifier Drug Interactions for ABI-H2158 in Healthy Adult Subjects
Brief Title: A Study to Assess CYP3A4 Modulator, Oral Contraceptive, and pH Modifier Drug Interactions for ABI-H2158 in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Assembly Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ABI-H2158-103
Record Dates: First submitted 2019-10-16; First posted 2019-10-29 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Itraconazole; Rifampin; Midazolam; Ethinyl Estradiol-Norgestrel Combination; Esomeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort 1: ABI-H2158 + Itraconazole (Experimental): Oral ABI-H2158 on Days 1 and 9; oral itraconazole once-daily (QD) on Days 6 through 13
  Interventions: Drug: ABI-H2158; Drug: Itraconazole
- Cohort 2: ABI-H2158 + Rifampin (Experimental): Oral ABI-H2158 on Days 1 and 12; oral rifampin QD on Days 6 through 16
  Interventions: Drug: ABI-H2158; Drug: Rifampin
- Cohort 3: ABI-H2158 + Esomeprazole (Experimental): Oral ABI-H2158 on Days 1 and 11; oral esomeprazole QD on Days 6 through 11
  Interventions: Drug: ABI-H2158; Drug: Esomeprazole
- Cohort 4: ABI-H2158 + Midazolam (Experimental): Oral midazolam on Days 1 and 11; oral ABI-H2158 QD on Days 2 through 11
  Interventions: Drug: ABI-H2158; Drug: Midazolam
- Cohort 5: ABI-H2158 + Oral Contraceptive (Experimental): Cycle 1: active oral contraceptive (ethinyl estradiol/levonorgestrel) QD on Days 1 through 21 and oral placebo QD on Days 22 through 28; Cycle 2: active oral contraceptive QD on Days 1 through 21, oral placebo QD on Days 22 through 26, and oral ABI-H2158 QD on Days 11 through 24
  Interventions: Drug: ABI-H2158; Drug: Ethinyl Estradiol / Levonorgestrel; Drug: Placebo matching oral contraceptive

INTERVENTIONS:
Drug: ABI-H2158 — ABI-H2158 tablets
Drug: Itraconazole — Itraconazole capsules
  Arms: Cohort 1: ABI-H2158 + Itraconazole
Drug: Rifampin — Rifampin capsules
  Arms: Cohort 2: ABI-H2158 + Rifampin
Drug: Midazolam — Midazolam syrup
  Arms: Cohort 4: ABI-H2158 + Midazolam
Drug: Ethinyl Estradiol / Levonorgestrel — Ethinyl Estradiol / Levonorgestrel tablets
  Arms: Cohort 5: ABI-H2158 + Oral Contraceptive
Drug: Esomeprazole — Esomeprazole capsules
  Arms: Cohort 3: ABI-H2158 + Esomeprazole
Drug: Placebo matching oral contraceptive — Placebo matching Ethinyl Estradiol / Levonorgestrel tablets
  Arms: Cohort 5: ABI-H2158 + Oral Contraceptive

SUMMARY:
This study is designed to assess 1) the effect of multiple doses of itraconazole (CYP3A4 inhibitor), rifampin (CYP3A4 inducer), and esomeprazole (pH modifier) on the pharmacokinetics of a single oral dose of ABI-H2158, and 2) the effect of steady-state oral ABI-H2158 on the pharmacokinetics of midazolam (sedative) and levonorgestrel/ethinyl estradiol (active oral contraceptive) in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

1. No clinically significant abnormal findings on physical exam, medical history, or clinical laboratory results at screening.
2. Cohort 5: naive to the use of oral contraceptives.

Exclusion Criteria:

1. Positive test results for human immunodeficiency virus (HIV) or hepatitis B or C.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-10-18 (Actual); Primary Completion 2020-01-12 (Actual); Study Completion 2020-01-29 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration time curve (AUC) of ABI-H2158 | before dosing and at pre-specified time points up to Day 17
Maximum observed plasma concentration (Cmax) of ABI-H2158 | before dosing and at pre-specified time points up to Day 17
AUC of Midazolam | before dosing and at pre-specified time points up to Day 12
Cmax of Midazolam | before dosing and at pre-specified time points up to Day 17
AUC of ethinyl estradiol and levonorgestrel | before dosing and at pre-specified time points up to 5 days after dosing on Day 21 of Cycle 1 and Cycle 2. Cycle 1 is 28 days and Cycle 2 is 26 days
Cmax of ethinyl estradiol and levonorgestrel | before dosing and at pre-specified time points up to 5 days after dosing on Day 21 of Cycle 1 and Cycle 2. Cycle 1 is 28 days and Cycle 2 is 26 days

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Study Lead, Study Director — Assembly Biosciences
Locations (1):
- Celerion, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: No